CLINICAL TRIAL: NCT03623750
Title: A Multicentre, Open-Label, Exploratory Phase Ib Clinical Study to Assess Safety and Efficacy of an EGFR Tyrosine Kinase Inhibitor in Combination With EGF Pathway Targeting Immunisation (EGF-PTI) in Treatment-Naïve Patients With EGFR Mutant NSCLC. The EPICAL Study
Brief Title: E GFR TKI and EGF-P TI C Ombination in EGFR mutA nt NSCL C
Acronym: EPICAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Oncológico Dr Rosell (Other)
Collaborators: Bioven Europe (Industry); MFAR (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MedOPP137; 2017-003237-28 (EudraCT Number)
Record Dates: First submitted 2018-07-20; First posted 2018-08-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: Open-label, uncontrolled, Phase Ib clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EGFR-TK Inhibitor plus EGF-PTI (Experimental): Elegile patients will receive a single pre-treatment low dose of intravenous cyclophosphamide 200mg/m2 before experimental treatment starts. Daily oral therapy with afatinib according to the SmPC of the product in nominal treatment cycles of 21 days followed by immunisation with EGF-PTI.
  Interventions: Drug: EGFR-TK Inhibitor; Biological: EGF-PTI; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: EGFR-TK Inhibitor — Patients will commence daily oral therapy with the EGFR TKI afatinib as soon as possible, preferably on the same day as low dose cyclophosphamide. Afatinib will be prescribed according to the Summary of Product Characteristics (SmPC) of the product, and will continue in nominal 21-day cycles for as long as clinically indicated.
Biological: EGF-PTI — The first day of dosing with EGF-PTI will be designated Day 1. Immunisation with EGF-PTI will commence 3 days after low dose cyclophosphamide and commencement of EGFR TKI, and will be repeated on Day 14, Day 28, Day 43, and Day 92. After the 5
  th vaccination, patients will enter a maintenance phase during which reduced dose vaccinations will be performed every 2 or 3 months in conjunction with the interval between detailed check-up of the patient. As this interval can vary between patients, the interval for maintenance vaccination can also vary between 2 and 3 months.
Drug: Cyclophosphamide — Eligible patients will receive a single pre-treatment of low dose of intravenous cyclophosphamide 200 mg/m2 (Day -3).

SUMMARY:
This is a multicentre, open-label, uncontrolled, Phase Ib clinical study. Patients who give informed consent will be screened for the study, including genotyping of the tumour and baseline characteristics. Eligible patients will receive a single pre-treatment of low dose of intravenous cyclophosphamide 200 mg/m2 (Day -3). Patients will commence daily oral therapy with the EGFR TKI afatinib as soon as possible, preferably on the same day as low dose cyclophosphamide. Afatinib will be prescribed according to the Summary of Product Characteristics (SmPC) of the product, and will continue in nominal 21-day cycles for as long as clinically indicated. The first day of dosing with EGF-PTI will be designated Day 1.

Immunisation with EGF-PTI will commence 3 days after low dose cyclophosphamide and commencement of EGFR TKI, and will be repeated on Day 14, Day 28, Day 43, and Day 92. After the 5 th vaccination, patients will be followed up every 6 weeks for basic safety data and every 3 months for complete efficacy data, safety data, and maintenance (reduced) doses of EGF-PTI. Patients will continue in the study until disease progression, death, safety concerns (in the opinion of the investigator), non-compliance with the protocol, the patient withdraws from the study, 1 year after randomisation of the last patient, or the study is stopped the sponsor, whichever occurs sooner

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Histological confirmation of locally advanced or metastatic, non-squamous NSCLC with an activating EGFR mutation who are not candidates for local curative treatment.
3. Stage IV, according to TNM Version 8, including M1a (malignant effusion) or M1b (distant metastasis), or locally advanced disease for which there is no curative treatment (including patients who progress after chemoradiotherapy in Stage III disease).
4. Centrally confirmed EGFR exon 19 deletion, exon 21 (L858R, L861Q) or exon 18 (G719X) mutation before treatment (concomitant T790M pre-treatment mutation is permitted).
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Existence of measurable or evaluable disease (according to RECIST 1.1 criteria). Patients with asymptomatic and stable brain metastases are eligible for the study.
7. Possibility of obtaining tissue samples, via a biopsy or surgical resection of the primary tumour or metastatic tumour tissue, within 60 days prior to the start of treatment.
8. Life expectancy ≥12 weeks.
9. Adequate haematological function, defined as: absolute neutrophil count (ANC) >1.5 x 109/L, platelet count >100.0 x 109/L, and haemoglobin >9.0 g/dL (>6.2 mmol/L).
10. Adequate coagulation, defined as: international normalised ratio (INR) ≤1.5.
11. Adequate liver function, defined as: total bilirubin <1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) <2.5 x ULN, alkaline phosphatase <5 ULN, except in the presence of single bone metastases and in the absence of any liver disorders.
12. Adequate renal function, defined as: calculated creatinine clearance >50 mL/min (Cockcroft-Gault formula) and proteinuria <2+ (dipstick).
13. Ability to complete the study, and residing within geographical proximity allowing for adequate follow-up.
14. Resolution of all acute toxic effects of any previous anti-cancer therapy (which can only be adjuvant or neoadjuvant) or previous surgical interventions not exceeding grade ≤1 according to the National Cancer Institute CTCAE Version 4.0 (except for alopecia or other side effects that the investigator does not consider to be a risk to patient safety).
15. All men, and women of childbearing potential, must agree to use a contraception method during the study treatment period and for at least 12 months after the last dose of EGF-TKI. Sexually active men, and women of childbearing potential, who are unwilling to use a contraceptive method are not eligible for the study.
16. Provision of written informed consent, signed and dated by the patient and the investigator, before any study interventions are performed.

Exclusion Criteria:

1. Locally advanced lung cancer candidate for curative treatment through radical surgery and/or radiotherapy, or chemotherapy.
2. Diagnosis with another lung cancer subtype, patients with mixed NSCLC with predominantly squamous cell cancer, or with any small-cell lung cancer component.
3. Presence or history of any other primary malignancy other than NSCLC within 5 years prior to enrolment into the study. Patients with a history of adequately treated basal or squamous cell carcinoma of the skin or any adequately treated in situ carcinoma may be included in the study.
4. Presence of one measurable or evaluable tumour lesion that has been resected or irradiated prior to enrolment in the study.
5. Receipt of prior antineoplastic treatment for advanced disease.
6. Prior treatment with cytotoxic chemotherapy for advanced NSCLC; neoadjuvant/adjuvant chemotherapy is permitted if at least 6 months have elapsed between the end of chemotherapy and the first day of EGF-PTI.
7. Previous treatment for lung cancer with an EGFR.
8. Concomitant use of immunosuppressant drugs such as azathioprine, tacrolimus, cyclosporine, etc. Use is not permitted within 1 month before screening.
9. Concomitant treatment with any other immunotherapy.
10. Receipt of other vaccines (with the exception of the influenza vaccine), within 1 month before screening.
11. Concomitant treatment with oral, intramuscular or intravenous corticosteroids. Use is not permitted within 1 month before screening. Inhaled corticosteroids to treat respiratory insufficiency (e.g. chronic obstructive pulmonary disease), or topical steroids are permitted.
12. Treatment with an investigational drug within 3 weeks before the first dose of EGF-PTI.
13. Patients of either sex who are unwilling to use an adequate contraception method until 12 months after the last dose of EGF-PTI or EGFR TKI, whichever is later.
14. History of interstitial lung disease induced by drugs, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active interstitial lung disease.
15. Any of the following ECG abnormalities:

    * Corrected QT interval (QTc) >470 msec, obtained from 3 ECGs at rest, using the QTc value determined according to the clinical screening ECG machine.
    * Any clinically significant abnormality in ECG rhythm, conduction or morphology at rest.
    * Any factor that increases the risk of QTc prolongation or risk of irregular heartbeat or sudden inexplicable death under the age of 40 in first-degree relatives or any concomitant medications that prolong the QT interval.
16. Uncontrolled, active or symptomatic metastases of the central nervous system (CNS), carcinomatous meningitis or leptomeningeal disease indicated by known clinical symptoms, cerebral oedema and/or progressive neoplasia. Patients with a history of CNS metastasis or compression of the spinal cord are eligible if they have received local final treatment (e.g., radiotherapy, stereotactic surgery) and if they have remained clinically stable without using anticonvulsants and corticosteroids for a minimum of 4 weeks prior to the first day of EGF-PTI treatment.
17. Patients who have had a surgical procedure unrelated to the study within 7 days prior to the first administration of EGF-PTI, or a significant traumatic lesion during the 4 weeks prior to starting the first dose of EGF-PTI, patients who have not recovered from the side effects of any major surgery or patients who might need major surgery during the course of the study.
18. Pregnant or breastfeeding women. Women of childbearing potential, including women who had their last menstrual period within the last 2 years, must have a negative serum or urine pregnancy test in the 7 days prior to the first dose of EGF-PTI.
19. Patients with a serious concomitant systemic disorder (e.g., active infection, including HIV or heart disease) that is incompatible with the study (in the opinion of the investigator), history of bleeding diathesis or anticoagulant therapy (the use of low molecular weight heparin is permitted provided that it is used for prophylaxis).
20. Treatment with any of the prohibited concomitant medications that cannot be stopped for the duration of trial participation.
21. Any other reason that the investigator deems to be incompatible with the patient's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of Adverse Events | 36 months
  Evaluate the safety and tolerability of epidermal growth factor receptor tyrosine kinase inhibitor plus EGF-PTI in newly diagnosed patients with advanced or metastatic non-squamous NSCLC with EGFR mutations who are not candidates for local curative treatment throughout the patient's participation in the study.

SECONDARY OUTCOMES:
Clinical response efficacy assessments | 36 months
  Evaluate the anti-tumor activity of epidermal growth factor receptor tyrosine kinase inhibitor plus EGF-PTI in terms of clinical response. Every 3 months after the first dose of EGF-PTI and throughout the patient's participation in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Andrés Aguilar Hernández, M.D., PhD., Study Director — Instituto Oncológico Dr Rosell; Andrés Aguilar Hernández, M.D., PhD., Study Chair — Instituto Oncológico Dr Rosell
Locations (4):
- Spain (4):
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Instituto Oncológico Dr. Rosell, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Universitario Regional de Málaga, Málaga

IPD SHARING:
Plan to Share IPD: No